CLINICAL TRIAL: NCT01770860
Title: An Assessment of QuiltVent™ Pad Technology on the Healing of Induced Dermabrasion Wounds
Brief Title: A Test of Different Kinds of Bandages on Healing of Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Products Company Division of Johnson & Johnson Consumer Companies, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: ABDWDP0005
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Wound Healing
Keywords: Adhesive Bandages; Dermabrasion Wounds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 6660 (Active Comparator): Five dermabrasion wounds will be created on each subject's back by a licensed physician. Four of the wounds will be covered with four different commercially-available bandages (6660, 4314, 8336 and 4840), and one wound will be left open to the air to serve as a no treatment control (0000). Treatments and control will be randomized to application site.
  Interventions: Device: 6660
- 4314 (Active Comparator): Five dermabrasion wounds will be created on each subject's back by a licensed physician. Four of the wounds will be covered with four different commercially-available bandages (6660, 4314, 8336 and 4840), and one wound will be left open to the air to serve as a no treatment control (0000). Treatments and control will be randomized to application site.
  Interventions: Device: 4314
- 8336 (Active Comparator): Five dermabrasion wounds will be created on each subject's back by a licensed physician. Four of the wounds will be covered with four different commercially-available bandages (6660, 4314, 8336 and 4840), and one wound will be left open to the air to serve as a no treatment control (0000). Treatments and control will be randomized to application site.
  Interventions: Device: 8336
- 4840 (Placebo Comparator): Five dermabrasion wounds will be created on each subject's back by a licensed physician. Four of the wounds will be covered with four different commercially-available bandages (6660, 4314, 8336 and 4840), and one wound will be left open to the air to serve as a no treatment control (0000). Treatments and control will be randomized to application site.
  Interventions: Device: 4840
- 0000 (No Intervention): Device: 0000
  At each daily visit, designated study personnel will cut out the center pad of the bandage and apply only the adhesive tabs around the assigned wound site.
  Other Names:
  * Sheer Strips
  * BAND-AID® with QuiltVent™ Pad Technology
  Five dermabrasion wounds will be created on each subject's back by a licensed physician. Four of the wounds will be covered with four different commercially-available bandages (6660, 4314, 8336 and 4840), and one wound will be left open to the air to serve as a no treatment control (0000). Treatments and control will be randomized to application site.

INTERVENTIONS:
Device: 6660 — At each daily visit, designated study personnel will replace the specific test product on the assigned wound site.
  Other Names: Sheer Strips; BAND-AID® with QuiltVent™ Pad Technology
  Arms: 6660
Device: 4314 — At each daily visit, designated study personnel will replace the specific test product on the assigned wound site.
  Other Names: Flexible Fabric; BAND-AID® with QuiltVent™ Pad Technology
  Arms: 4314
Device: 8336 — At each daily visit, designated study personnel will replace the specific test product on the assigned wound site.
  Other Names: Tough Strips® Waterproof; BAND-AID® with QuiltVent™ Pad Technology
  Arms: 8336
Device: 4840 — At each daily visit, designated study personnel will replace the specific test product on the assigned wound site.
  Other Names: Flat Pad; BAND-AID® Dora the Explorer™
  Arms: 4840

SUMMARY:
This two-week study will compare the healing of minor wounds when no bandage is applied against four different types of bandages.

The study investigators will make five small wounds similar to scrapes (about a half-inch square) on the back of subjects who qualify to participate in the trial and have given informed consent. Four of the wounds will be covered by different bandages and one will be left uncovered. Participants will visit the clinic every day for 2 weeks or until all the wounds are healed (whichever comes first). At the clinic, the bandages will be removed, the doctor will score the wounds, a picture will be taken of the wounds and new bandages will be applied.

It is expected that some pain and itching will be experienced, because they are part of the normal wound healing process. Subjects will be asked about adverse events at each visit and will have the opportunity to discuss issues or concerns with the investigator or the doctor during the course of the trial. It is expected that the wounds will be completely healed within 14 days, but if not, the participant will need to return to the clinic for follow-up treatment until the wounds are completely healed.

We will see if the different bandages help with the healing of the wounds during the study.

DETAILED DESCRIPTION:
This study is evaluating the performance of various bandages on facilitating the healing of induced dermabrasion wounds. To qualify for this study, subjects must meet the inclusion/exclusion criteria within the protocol-specified parameters at both the screening and baseline visits. Once a subject is qualified, five dermabrasion wounds will be created on each subject's back by a licensed physician. Four of the wounds will be covered with four different commercially-available bandages and one wound will be left open to the air to serve as a no treatment control. Treatments and control will be randomized to application site. During this 14-day clinical study, subjects will return to the site for daily evaluations; study bandages will also be replaced daily by study personnel. Adverse events will be observed and collected by querying each subject at each visit, and during any follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to read and understand English enough to understand the nature, risk and relevance of the study, read and sign the informed consent document, and follow study instructions
* After being completely informed about the study and being given a chance to have all questions answered, the subject has signed an informed consent document agreeing to:
* comply with lifestyle instructions, including: limiting bandage exposure to water or sunlight, the use of lotions, creams, cosmetics or sunscreens during the study, to allow at least 2 hours between showers and scheduled visits, and the use of contraception
* return to the clinical site for follow-up visits if the wounds are not healed by Day 14
* Subject is determined to be an appropriate participant according to protocol-defined conditions, including among other things, Body Weight and Fitzpatrick Skin Type between I (Always burns easily, never tans) and III (Burns moderately, tans gradually)
* In the opinion of the Investigator, participation in the trial will not compromise the subject's safety or the interpretation of study results

Exclusion Criteria:

* Medical condition or history, or use of drugs or treatments that could possibly compromise the safety of the research subject or the interpretation of results, per protocol or in the opinion of the investigator
* Known allergies or hypersensitivity to LATEX, anesthetics, adhesive bandages, wound treatment products or any component present in the test bandages
* Current participation in any other clinical trial or past participation in other clinical trials described in the protocol
* Body mass index (BMI) above 35, and/or Fitzpatrick Skin Type above III
* Pregnant, nursing or planning a pregnancy

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Kendall, Study Director — Johnson & Johnson Consumer Products Company Division of Johnson & Johnson Consumer Companies, Inc.
Locations (1):
- Hill Top Research, St. Petersburg, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One additional subject was enrolled but withdrew before randomization.
Groups:
- 4 Commercially-available Bandage and 1 Control: Five dermabrasion wounds will be created on each subject's back by a licensed physician. Four of the wounds will be covered with four different commercially-available bandages (6660, 4314, 8336 and 4840), and one wound will be left open to the air to serve as a no treatment control (0000). Treatments and control will be randomized to application site.
Period: Overall Study
Arm/Group | 4 Commercially-available Bandage and 1 Control
Started | 46 (Forty-six subjects were enrolled but one subject withdrew before randomization.)
Randomization | 45 (One participant withdrew before randomization)
Completed | 40
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Not completed — Administrative decision made by the PI | 1

BASELINE CHARACTERISTICS:
Arm/Group | 4 Commercially-available Bandage and 1 Control
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (7.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45
Fitzpatrick Skin Classification [Number; unit: participants] — The Fitzpatrick skin classification is based on the skin's unprotected response to the first 30-45 minutes of sun exposure after a winter season without sun exposure. The classification is on a scale from I to VI where I = always burns easily; never tans and VI =Never burns; deeply pigmented.
  participants
    Fitzpatrick Skin Classification - II | 11
    Fitzpatrick Skin Classification - III | 34

OUTCOME MEASURES:

1. Primary Outcome: Time to Healing (Days)
Description: Wound epithelialization will be recorded daily for each wound (until healed) by the doctor on a scale of 0-5, where 0= No presence of epithelialization (no sign of healing), a bandage is necessary and 5=Wound is 100% epithelialized (healed), no bandage necessary. The median time to healing will be estimated from the survival curves using the Kaplan-Meier method for each test product. Time to healing is defined as the time from wounding to 12:00 pm of the day the wound is 100% epithelialized (receives a score of 5). If the wound is not 100% epithelialized on Day 14 or on the last day of visit, Time to healing will be considered as censored.
Time Frame: within 14 days
Population: The Intent-to-Treat (ITT) population is defined as all subjects who received study bandages. Forty six subjects were enrolled but one withdrew before randomization.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Bandage QuiltVent™ Sheer Strips (With Pad Removed): No treatment
Arm/Group | Bandage QuiltVent™ Sheer Strips (With Pad Removed) | Bandage QuiltVent™ Sheer Strips | Bandage QuiltVent™ Flexible Fabric | Bandage QuiltVent™ Tough Strips Waterproof | Bandage Dora the Explorer™
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 45
days | 13.1 [12.95 to 13.14] | NA [NA to NA] — Due to the censoring status of the data, the median time to healing could not be estimated | 13.1 [13.05 to 13.15] | NA [10.90 to NA] — Due to the censoring status of the data, the median time to healing could not be estimated | NA [NA to NA] — Due to the censoring status of the data, the median time to healing could not be estimated

2. Secondary Outcome: Forced Rank Score
Description: The wound evaluator will rank the overall appearance of all five wounds in relation to each other on a daily basis until all five are healed on a scale of 1 to 5, where 1= Worst and 5=Best. The forced Rank was evaluated at each visit. The mean score derived as total score divided by visit number 13 was analyzed using a mixed model.
Time Frame: within 14 days
Population: The Intent-to-Treat (ITT) population is defined as all subjects who received study bandages. One randomized subject withdrew from the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bandage QuiltVent™ Sheer Strips (With Pad Removed) | Bandage QuiltVent™ Sheer Strips | Bandage QuiltVent™ Flexible Fabric | Bandage QuiltVent™ Tough Strips Waterproof | Bandage Dora the Explorer™
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 44
scores on a scale | 1.48 (0.58) [NA to NA] | 3.04 (0.90) [1.24 to 1.88] | 2.44 (0.95) [0.65 to 1.28] | 3.77 (1.01) [1.97 to 2.61] | 3.29 (0.95) [1.50 to 2.13]
Statistical Analysis 1: Comparison: Bandage QuiltVent™ Sheer Strips (With Pad Removed) vs Bandage QuiltVent™ Sheer Strips vs Bandage QuiltVent™ Flexible Fabric vs Bandage QuiltVent™ Tough Strips Waterproof vs Bandage Dora the Explorer™; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The p-values presented were for each of the bandage groups compared to no treatment group; P-value is from mixed model with Treatment (trt) as fix effect, and subject as random effect

3. Secondary Outcome: Erythema
Description: Until healed, erythema (redness) of each wound bed and surrounding skin will be scored daily on a scale of 0-10, where 0=None and 10=Most severe. Erythema was evaluated at each visit. The mean score derived as total score divided by visit number 13 was analyzed here using a mixed model.
Time Frame: within 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bandage QuiltVent™ Sheer Strips (With Pad Removed) | Bandage QuiltVent™ Sheer Strips | Bandage QuiltVent™ Flexible Fabric | Bandage QuiltVent™ Tough Strips Waterproof | Bandage Dora the Explorer™
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 44
scores on a scale | 1.74 (0.64) [NA to NA] | 0.90 (0.42) [-1.02 to -0.67] | 0.90 (0.49) [-1.01 to -0.66] | 0.97 (0.48) [-0.94 to -0.59] | 0.88 (0.43) [-1.03 to -0.68]
Statistical Analysis 1: Comparison: Bandage QuiltVent™ Sheer Strips (With Pad Removed) vs Bandage QuiltVent™ Sheer Strips vs Bandage QuiltVent™ Flexible Fabric vs Bandage QuiltVent™ Tough Strips Waterproof vs Bandage Dora the Explorer™; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The p-values presented were for each of the bandage groups compared to no treatment group; P-value is from mixed model with treatment (trt) as fix effect, and subject as random effect

4. Secondary Outcome: Edema
Description: Until healed, edema (swelling) of each wound bed and surrounding skin will be scored daily on a scale of 0-10, where 0=None and 10=Most severe. Mean Edema was evaluated at each visit. The mean score derived as total score divided by visit number 13 was analyzed using a mixed model.
Time Frame: within 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bandage QuiltVent™ Sheer Strips (With Pad Removed) | Bandage QuiltVent™ Sheer Strips | Bandage QuiltVent™ Flexible Fabric | Bandage QuiltVent™ Tough Strips Waterproof | Bandage Dora the Explorer™
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 44
scores on a scale | 1.44 (0.52) | 0.57 (0.38) | 0.69 (0.43) | 0.56 (0.42) | 0.64 (0.39)
Statistical Analysis 1: Comparison: Bandage QuiltVent™ Sheer Strips (With Pad Removed) vs Bandage QuiltVent™ Sheer Strips vs Bandage QuiltVent™ Flexible Fabric vs Bandage QuiltVent™ Tough Strips Waterproof vs Bandage Dora the Explorer™; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The p-values presented were for each of the bandage groups compared to no treatment group; P-value is from mixed model with treatment (trt) as fix effect, and subject as random effect

5. Secondary Outcome: Maceration
Description: Until healed, maceration (a slight whitening of the skin around the wound compared to the surrounding unbandaged area) will be scored as P=Present or A=Absent. Percentage of maceration was derived as the maceration presence times over study period divided by visit number 13.
Time Frame: within 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of maceration
Arm/Group | Bandage QuiltVent™ Sheer Strips (With Pad Removed) | Bandage QuiltVent™ Sheer Strips | Bandage QuiltVent™ Flexible Fabric | Bandage QuiltVent™ Tough Strips Waterproof | Bandage Dora the Explorer™
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 44
percentage of maceration | 4.37 (9.15) | 70.98 (22.12) | 65.21 (23.43) | 39.34 (31.88) | 63.99 (26.64)
Statistical Analysis 1: Comparison: Bandage QuiltVent™ Sheer Strips (With Pad Removed) vs Bandage QuiltVent™ Sheer Strips vs Bandage QuiltVent™ Flexible Fabric vs Bandage QuiltVent™ Tough Strips Waterproof vs Bandage Dora the Explorer™; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The p-values presented were for each of the bandage groups compared to no treatment group; P-value is from mixed model with treatment (trt) as fix effect, and subject as random effect

6. Secondary Outcome: Subjective Assessment of Pain
Description: Until healed, pain assessments by the participant will be recorded daily for each wound site as either Present (P) or Absent (A). Percentage of pain was derived as the pain presence times over study period divided by visit number 13.
Time Frame: within 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of pain
Arm/Group | Bandage QuiltVent™ Sheer Strips (With Pad Removed) | Bandage QuiltVent™ Sheer Strips | Bandage QuiltVent™ Flexible Fabric | Bandage QuiltVent™ Tough Strips Waterproof | Bandage Dora the Explorer™
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 44
percentage of pain | 5.24 (12.39) | 4.55 (10.13) | 2.45 (6.38) | 3.85 (7.87) | 2.45 (5.69)
Statistical Analysis 1: Comparison: Bandage QuiltVent™ Sheer Strips (With Pad Removed) vs Bandage QuiltVent™ Sheer Strips vs Bandage QuiltVent™ Flexible Fabric vs Bandage QuiltVent™ Tough Strips Waterproof vs Bandage Dora the Explorer™; Test type: Superiority or Other; p = 0.0476, Mixed Models Analysis; P-value is from mixed model with treatment (trt) as fix effect, and subject as random effect

7. Secondary Outcome: Subjective Assessment of Itch
Description: Until healed, itch assessments by the participant will be recorded daily for each wound site as either Present (P) or Absent (A). Percentage of itch was derived as the itch presence times over study period divided by visit number 13.
Time Frame: within 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of itching
Arm/Group | Bandage QuiltVent™ Sheer Strips (With Pad Removed) | Bandage QuiltVent™ Sheer Strips | Bandage QuiltVent™ Flexible Fabric | Bandage QuiltVent™ Tough Strips Waterproof | Bandage Dora the Explorer™
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 44
percentage of itching | 21.33 (28.24) | 26.22 (29.46) | 16.43 (21.73) | 25.87 (26.24) | 20.10 (22.15)

8. Secondary Outcome: Subjective Assessment of Wound Healing
Description: Until healed, subjects will be shown photographs of each wound they have not previously classified as healed at each daily visit, and asked to determine if the wound is healed. Yes or No responses will be recorded, along with text entries of the reasons for the response. This outcome measure reports the number of subjects who report that the wound has healed.
Time Frame: within 14 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Bandage QuiltVent™ Sheer Strips (With Pad Removed) | Bandage QuiltVent™ Sheer Strips | Bandage QuiltVent™ Flexible Fabric | Bandage QuiltVent™ Tough Strips Waterproof | Bandage Dora the Explorer™
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 44
Participants | 22 | 20 | 14 | 30 | 26

ADVERSE EVENTS:
Time Frame: 30 days and beyond for serious adverse events if assessed as possibly treatment related. Visits 2-15 and beyond if needed for adverse events.
Description: The safety population was 46. One subject withdrew from the study, before randomization or receving treatment, due to a serious adverse event.
  Adverse events were collected for all five interventions simultaneously without attributing causal relationship to a particular intervention.
Arm/Group | 4 Commercially-available Bandage and 1 Control
Serious Adverse Events (participants affected / at risk) | 1/46
Other Adverse Events (participants affected / at risk) | 11/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 Commercially-available Bandage and 1 Control (N=46)
Bronchopneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 Commercially-available Bandage and 1 Control (N=46)
Headache (Nervous system disorders) | 6
Excoriation (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Tooth Abscess (Infections and infestations) | 1
Influenza Like Illness (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days